CLINICAL TRIAL: NCT03700008
Title: Development of a Digital Content-free Speech Analysis for the Measurement of Mental Health and Follow-up of Mental Disorders
Brief Title: Content-free Speech Analysis for Measurement of Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuropsychiatrischen Zentrums Hamburg-Altona (Other)
Collaborators: VoiceSense Ltd. Herzelba, Israel (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TONN_2018_01
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Mental Disorder; Conditions Influencing Health Status
Keywords: Mental Disorder; Treatment planning; Technical measurements of mental state; Course-prediction of Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Two randomized groups of participants, blinded to rater in relation of the diagnosis of the individual proband.
Who Masked: Outcomes Assessor
Masking Description: The outcome-assessor or rater did not know which diagnosis the participant has and the participant is informed about the diagnosis after the diagnostic procedure from a physician/ psychotherapist not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with mental illness (Other): Participant with pre known or actually diagnosed mental disorder, especially affective or neurodevelopmental disorder.
  Using the speech analysis tool with 120 seconds of free speech, measure the mental state with SCL-90, PRIME-MD, B5T, ADHD-VAS as conventional psychological measurements.
  Interventions: Diagnostic Test: Speech analysis tool; Diagnostic Test: Conventional psychological measurements
- Participants without any mental illness (Other): Participant with never diagnosed mental disorder, in a healthy mental state. Using the speech analysis tool with 120 seconds of free speech, measure the mental state with SCL-90, PRIME-MD, B5T, ADHD-VAS as conventional psychological measurements.
  Interventions: Diagnostic Test: Speech analysis tool; Diagnostic Test: Conventional psychological measurements

INTERVENTIONS:
Diagnostic Test: Speech analysis tool — Using the speech analysis tool with recording 120 seconds of free speech and analysis of 200 content-free parameters of the speech including factor analytic process to compress the data to 5-10 core parameters.
Diagnostic Test: Conventional psychological measurements — Using well known and validated psychological measurements to identify the mental state of the participants.

SUMMARY:
Trial to prove the functionality and efficacy of a content-free speech analysis tool to detect problematic mental health status or phases of patients with pre known or unknown mental health disorders, focussed on affective disorders or neurodevelopmental disorders. The participants talk in free speech to the tool, this will be analyzed content-free and compared with psychological instruments to detect the mental status in conventional way.

DETAILED DESCRIPTION:
Participants with and without pre known mental disorders will be recruited and analyzed with speech analysis and conventional psychological instruments, as primary measurement the SCL-90-Scale, as secondary instruments the PRIME-MD (explicit in use the PHQ-9 for depressive symptoms and the GAD-7 for anxiety), B5T and an ADHD-VAS-Score (t0). Then the investigators check the status of the participants later at t1 (4-6 weeks after t0) and t2 (4-6 weeks after t1).

The speech measuring instruments is the "VoiceSense" digital voice analysis tool, which enables the analysis of 200 specific speech parameters and the assessment of the findings through the use of psychometric instruments and questionnaires.

The hypothesis is that the data of the voicesense analysis tool compared to the psychological instruments provide a good match and the voicesense technique can be used as a predictive and course-description tool in mental illness.

ELIGIBILITY:
Inclusion Criteria:

* being regular outpatient with mental disorder (verum group)
* being voluntary participant without mental disorder (control group)
* native german language speakers
* in good general health (absence of cancer, acute myocardial infarction, unstable angina, severe cardiac arrhythmia, recent cerebrovascular incident, or severe atherosclerosis)

Exclusion Criteria:

* schizophrenia
* dementia
* pregnancy or breastfeeding
* current or recent (less than 1 year) history of alcohol and/or drug abuse
* current or recent (less than 1 year) history of suicide attempts
* other significant comorbidities according to the Investigator's clinical assessment (for example, cancer, acute myocardial infarction, unstable angina, severe cardiac arrhythmia, recent cerebrovascular incident, or severe atherosclerosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Global scores of Symptom-Checklist 90 (SCL-90) | score at the date of start of participation (day 1)
  The SCL-90 evaluates the psychological distress during the past seven days using nine scales for primary symptom dimensions and three scores among global distress indices. The basic psychological distress is determined by the GSI (Global Severity Index), the intensity of the responses by the PSDI (Positive Symptom Distress Index) and by the PST (Positive Symptom Total). The global scales provide an overview of the severity of the psychological distress. The scores ranged from 0.0 to 2.9 (GSI), 0-90 (PSI) and 0.0-2.9 (PSDI), all were calculated in T-values, so no cut-off but reliable T-values are published.

SECONDARY OUTCOMES:
Global score of depression measured with the "Patients-Health-Questionnaire 9" (PHQ9) | score at the date of start of participation (day 1)
  The PHQ-9 is a diagnostic tool, extracted from the PRIME-MD of Spitzer et al., used in DSM-5-diagnostic criteria for defining major depressive disorder. There is a Range from 9 to 36, the cut off for diagnosis of depressive disorder is 15
Global score of anxiety, measured with the "Generalized Anxiety Disorder 7" GAD-7 | score at the date of start of participation (day 1)
  The GAD-7 is a diagnostic tool, extracted from the PRIME-MD of Spitzer et al., used in many studies and clinical practice to identify anxiety disorders. There is a Range from 7 to 21, the cut off for diagnosis of anxiety disorder is 9 (cutoff score 10-> sensitivity 89%, specificity 82%, test-retest reliability with ICC=0.83)
Personality disorders and states, measured with the Big five personality test (B5T) | score at the date of start of participation (day 1)
  The B5T is a diagnostic tool to measure the impact of personality traits extraversion, consciousness, neuroticism, openess, agreeableness and three special motivational scales. There are 72 items, the overall-consistency is good, the test is evaluated in a german population sample with N= 7400.
Visuel analogue scale Attention-Deficit-Hyperactivity-Disorder (ADHD-VAS) | score at the date of start of participation ("day 1")
  The ADHD-VAS is a compressed form to ask the three core-parameters of ADHD in participants with diagnosed adult ADHD, hyperactivity, impulsivity/emotional stability and inattention. There are three visual scores, ranges from 0 to 10 each, cut-off is 4 each.
Changes of global scores of Symptom-Checklist 90 (SCL-90) | scores an average 5 weeks after day 1 and changes compared to scores at day 1
  The SCL-90 evaluates the psychological distress during the past seven days using nine scales for primary symptom dimensions and three scores among global distress indices. The basic psychological distress is determined by the GSI (Global Severity Index), the intensity of the responses by the PSDI (Positive Symptom Distress Index) and by the PST (Positive Symptom Total). The global scales provide an overview of the severity of the psychological distress. The scores ranged from 0.0 to 2.9 (GSI), 0-90 (PSI) and 0.0-2.9 (PSDI), all were calculated in T-values, so no cut-off but reliable T-values are published.
Changes of global scores of Symptom-Checklist 90 (SCL-90) | scores at an average 10 weeks after day 1 and changes compared to scores at day 1
  The SCL-90 evaluates the psychological distress during the past seven days using nine scales for primary symptom dimensions and three scores among global distress indices. The basic psychological distress is determined by the GSI (Global Severity Index), the intensity of the responses by the PSDI (Positive Symptom Distress Index) and by the PST (Positive Symptom Total). The global scales provide an overview of the severity of the psychological distress. The scores ranged from 0.0 to 2.9 (GSI), 0-90 (PSI) and 0.0-2.9 (PSDI), all were calculated in T-values, so no cut-off but reliable T-values are published.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Tonn, MD, Principal Investigator — Director
Locations (1):
- Neuropsychiatric Center of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tonn P, Seule L, Degani Y, Herzinger S, Klein A, Schulze N. Digital Content-Free Speech Analysis Tool to Measure Affective Distress in Mental Health: Evaluation Study. JMIR Form Res. 2022 Aug 30;6(8):e37061. doi: 10.2196/37061. PMID 36040767
- [Derived] Tonn P, Degani Y, Hershko S, Klein A, Seule L, Schulze N. Development of a Digital Content-Free Speech Analysis Tool for the Measurement of Mental Health and Follow-Up for Mental Disorders: Protocol for a Case-Control Study. JMIR Res Protoc. 2020 May 14;9(5):e13852. doi: 10.2196/13852. PMID 32406862